CLINICAL TRIAL: NCT04939883
Title: A Prospective Multi-Center Randomized Study to Evaluate the Effects of Carvedilol on Cardiotoxicity in Cancer Patients Submitted to Anthracycline Therapy
Brief Title: Effects of Carvedilol on Cardiotoxicity in Cancer Patients Submitted to Anthracycline Therapy
Acronym: CardioTox
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AVAP-NG 989
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Carvedilol; Anthracyclines; Cardiotoxicity; Chemotherapy
MeSH Terms: conditions — Neoplasms; Cardiotoxicity | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization will be in the proportion of 1: 1 (carvedilol x placebo). Both randomization and allocation of patients will be chosen in a veiled manner to patients and to assess. Data on randomization and allocation will be under custody of the Data analysis and safety committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Patients allocated to the intervention group will receive carvedilol 6.25 mg twice daily, then increased to 12.5 mg twice daily, until maximum dose of 25 mg twice daily according to the patients' tolerance; The dosis increments will occur every 5 days. If after the increment the patient develops bradycardia or hypotension, the dose will be reduced to the maximum tolerated dose. Carvedilol will ideally be maintained for up to 30 days after the end of chemotherapy.
  Interventions: Drug: Carvedilol
- Control Group (Placebo Comparator): Patients allocated to this group will receive placebo in a presumably staggered and progressive manner similar to the group intervention. The placebo will ideally be maintained for up to 30 days after the end of chemotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol — Carvedilol will be dispensed in a staggered and progressive manner, initially from 6.25 mg twice daily, then increased to 12.5 mg twice daily, until maximum dose of 25 mg twice daily or development of contraindications
  Arms: Intervention Group
Drug: Placebo — Patients will receive placebo in a presumed staggered and progressive manner similar to the intervention group. The placebo will ideally be maintained for up to 30 days after the end of chemotherapy.
  Arms: Control Group

SUMMARY:
Neoplasia is the main cause of general death in the Brazilian population. In 2016, they were responsible for approximately 211,343 (16%) deaths, followed by cardiovascular diseases (12.6%). Despite the high mortality rate of neoplasia, oncological treatment have advanced substantially in recent decades improving the prognosis of patients. However, growing evidence suggest that some oncological agents may induce significant toxicity that may play a major role in the quality of life, morbidity and mortality. The cardiovascular system is often negatively affected with cancer therapy, predisposing several patients to stop appropriate treatments or to have cardiovascular events related to the cardiotoxicity. The most typical manifestation of cardiotoxicity and related consequences (heart failure) are related to the use of anthracyclines. Anthracyclines are part of the chemotherapy regimen for solid tumors and hematological neoplasms in children and adults, and are associated with an increase in life expectancy. Carvedilol is an α and β-blocker that also has antioxidant properties. Preliminary studies have shown that carvedilol and its metabolites prevent lipid peroxidation, inhibit the formation and inactivate free radicals, in addition to preventing the depletion of endogenous antioxidants, such as vitamin E. These effects would potentially prevent anthracycline injury but definitive evidence is still needed. This is a multi-center, double-blind, randomized, placebo-controlled study that aims to establish the efficacy of carvedilol for the primary prevention of left ventricular systolic dysfunction in cancer patients obtained with anthracycline chemotherapy, in different schedules and doses.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of screening
* Cancer patients that will receive chemotherapy with anthracyclines.

Exclusion Criteria:

* Inability to adequate asses left ventricular function
* Previous symptoms (dyspnea on exertion, orthopnea, paroxysmal nocturnal dyspnea, and pulmonary and systemic congestion) suggestive of or a previous diagnosis of heart failure.
* Previous history of any cardiomyopathy (eg.: valve disease, Chagas' disease, infiltrative cardiomyopathy)
* LVEF < 50%
* Previous history of myocardial revascularization
* Permanent tachyarrhythmia (flutter, atrial fibrillation, atrial tachycardia)
* Congenital heart disease with left ventricular function impared
* Contra-indication to the use of beta-blockers.
* Pregnant or Breast-feeding females or women of childbearing age who intend to became pregnant.
* On kidney replacement therapy
* ECOG >= 4 or Karnofsky <=30
* Advanced hepatic failure (C score Child-Pugh and MELD > 15);
* Previous use of anthracycline
* Have any serious concomitant systemic disease, condition, or disorder that, in the opinion of the investigator, should preclude participation in this study
* Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1018 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Drop in ejection fraction within 12 months of starting treatment. | 12 months
  Drop in ejection fraction> 10% to values less than 50% of the left ventricle
Cardiac events within 12 months of starting treatment. | 12 months
  Cardiac events such as death, resuscitated cardiac arrest, myocardial infarction, heart failure and cardiac arrhythmias

SECONDARY OUTCOMES:
Drop in ejection fraction within 12 months. | 12 months
  Drop in ejection fraction greater than 10% and values less than 55%
Reduction in myocardial strain in 12 months from the start of treatment. | 12 months
  Relative reduction of more than 15% in myocardial strain
Diastolic dysfunction within 12 months | 12 months
  Development of diastolic dysfunction within 12 months
Elevation of biomarkers during chemotherapy and up to 12 months of follow-up | 12 months
  Elevation of biomarkers (NT-pro BNP and troponin) during chemotherapy and up to 24 months of follow-up
Quality of life (EuroQol-5D). | 12 months
  Quality of life measured by questionnaire in up to 12 months.
Cardiovascular complications in 12 months. | 12 months
  Cardiovascular complications (death, resuscitated cardiac arrest, myocardial infarction, heart failure and cardiac arrhythmias) in 24 months.

OTHER OUTCOMES:
Diagnosis of neoplasia within 12 months. | 12 months
  Diagnosis of another neoplasia
Progression of oncological disease within 12 months. | 12 months
  Progression of oncological disease
Tumor recurrence within 12 months. | 12 months.
  Tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Renato H D. lopes, MD, PhD, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospital Sirio Libanes, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa IBSDS, Furtado RHM, Drager LF, de Barros E Silva PGM, Melo MDT, Araruna P, Bacchiega BC, Cauduro S, Walter E, Fialho GL, Silvestre O, Damiani LP, Barbosa LM, Luz MN, Silva ACA, de Mattos RR, Saretta R, Rehder MHHS, Hajjar LA, Lopes-Fernandez T, Dent S, Gibson CM, Lopes RD, Kalil Filho R; on behalf the CARDIOTOX Investigators. Effects of carvedilol on the prevention of cardiotoxicity induced by anthracyclines: Design and rationale of the CARDIOTOX trial. Am Heart J. 2025 Jul;285:1-11. doi: 10.1016/j.ahj.2025.02.014. Epub 2025 Feb 22. PMID 39988204